CLINICAL TRIAL: NCT01668654
Title: RTG113388, a Long-term, Open-label Safety Extension Study of Retigabine/Ezogabine in Pediatric Subjects With Partial Onset Seizures (>= 12 Years Old) and Subjects With Lennox-Gastaut Syndrome (>=12 Years Old)
Brief Title: Long-term, Open-label Safety Extension Study of Retigabine/Ezogabine in Pediatric Subjects (>= 12 Years Old) With POS or LGS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA placed a clinical hold on the Pediatric Program requiring retigabine discontinuation in subjects; early termination allows for timely reporting of results.
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113388
Record Dates: First submitted 2012-05-17; First posted 2012-08-20 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Epilepsy
Keywords: Epilepsy; Partial Onset epilepsy; Lennox-Gastaut Syndrome; Open-label extension study
MeSH Terms: conditions — Epilepsy; Lennox Gastaut Syndrome | interventions — ezogabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- retigabine/ezogabine (Experimental): retigabine/ezogabine will be administered three times a day (TID) as add-on therapy based on weight
  Interventions: Drug: retigabine/ezogabine

INTERVENTIONS:
Drug: retigabine/ezogabine — retigabine/ezogabine will be administered three times a day (TID) as add-on therapy based on weight

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of retigabine/ezogabine as an adjunctive treatment in subjects with either partial onset seizures (12 to < 18 years old) or Lennox-Gastaut Syndrome (12 to <30 years old) who have participated in a previous ("parent") study.

DETAILED DESCRIPTION:
Epilepsy is among the most common serious neurologic disorders in childhood. Medicines with novel actions of mechanisms of action are needed to try to address the unmet clinical need for seizure control in patients with treatment-resistant epilepsy. The purpose of this study is to evaluate the long-term safety and tolerability of retigabine/ezogabine as an adjunctive treatment in subjects with either partial onset seizures (12 to < 18 years old) or Lennox-Gastaut Syndrome (12 to <30 years old) who have participated in a previous ("parent") study.

ELIGIBILITY:
Inclusion Criteria:

* Has participated in either a Phase II or Phase III retigabine/ezogabine clinical trial evaluating partial onset seizures or seizures comprising Lennox-Gastaut syndrome and met the requirements defined in the parent study to transition into the open-label extension study
* Investigator and caregiver consider it beneficial for the patient to continue treatment with retigabine/ezogabine
* Female subjects of child-bearing potential (after menarche) must either not be sexually active or must be practicing an acceptable method of contraception (documented in the medical chart) from two weeks prior to administration of study medication and for 28 days after completion or premature discontinuation from the study
* Subject is living with his/her custodial parent(s) or legal guardian(s) and has contact with them on a daily basis
* Written informed consent is obtained from the subjects parent/guardian and accompanying assent from subject. The subject, and/or his/her custodial parents(s) or legal guardian(s) have the ability to comprehend the key components of the informed consent form

Exclusion Criteria:

* Has insufficient ability to articulate the presence or absence of urinary tract symptoms
* Has experienced an adverse event, clinically significant laboratory abnormality or was discontinued from the parent study due to a reason that in the investigator's judgment would preclude enrollment to the study
* Has a urine sample with: Urine specific gravity >1.035, Urine pH <4.6 or >8.0, ≥2+ proteinuria, Casts or crystals (any type), >5 RBC/HPF, unrelated to menses
* Has a blood sample with: BUN >21 mg/dl for 12 year old, or >25 mg/dl for >12 year old, Creatinine >1.03 mg/dl (F), or >1.3 mg/dl (M), Uric acid >7.5 mg/dl (F), or >8.5 mg/dl (M), Chloride >108 mEq/L, parameters for calcium, inorganic phosphorous or CO2 that are clinically significant as judged by the investigator
* Has presence of clinically significant hepatic laboratory values: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >2x upper limit of normal (ULN); alkaline phosphatase and bilirubin ≥1.5xULN (isolated bilirubin >1.5ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%
* Has presence of clinically significant cardiac arrhythmias
* Has any abnormality on 12-lead ECG which is clinically significant in the opinion of the investigator, or has a corrected QT interval (using either Bazett's or Fridericia's) >500msec ( >530 msec for subjects with Bundle Branch Block), uncorrected QT interval >600msec, or change from baseline QTc >60msec
* Has a history of one or more renal calculi
* Has disturbances of micturition or known urinary obstructions, including renal calculi
* Has a documented anatomical stricture or other anatomical abnormality of the urinary tract system that has the potential to interfere with urinary flow
* Has experienced clinically significant urinary retention and/or required urinary catheterization in the preceding 6 months
* Has experienced 2 or more objectively documented urinary tract infections in the preceding 12 months
* Has a history of inadequate fluid intake and clinically significant dehydration in the preceding 6 months
* Within the preceding month, has taken anti-cholinergic medication on an ongoing basis
* Has active suicidal plan/intent or has had active suicidal thoughts in the past 6 months or has history of suicide attempt in the last 2 years or more than one lifetime suicide attempt
* Is planning surgery or implantation of a vagus nerve stimulator to control seizures during the study
* Is currently or has been abusing substance(s) or any medications in the 12 months prior to study entry
* Has taken an investigational drug (exception retigabine/ezogabine), or used an investigational device, within the previous 30 days prior, or plans to take an investigational drug anytime during the study
* Females who are lactating or are pregnant
* Unwillingness or inability to follow the procedures outlined in the protocol
* The subject is felt, by the investigator, to be unsuitable for inclusion in the study
* Children in care

Ages: 12 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2012-09-04 (Actual); Primary Completion 2013-06-18 (Actual); Study Completion 2013-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Wellington, Florida
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par.) aged 12 years or older, who had participated in a previous parent study GSK113284 (NCT014945840) evaluating Retigabine/Ezogabine in the treatment of partial onset seizures or seizures comprising Lennox-Gastaut syndrome, were enrolled in this open-label extension study.
Pre-assignment Details: Eligible par. began the Treatment Period at the eligibility assessment Visit followed by a 3-week Taper Phase, and a Follow-Up Visit within 3 days from the end of the Taper Phase. The study was prematurely discontinued after enrolling only 4 of the planned 500 par.
Groups:
- Retigabine/Ezogabine TID: Participants (par.) received retigabine/ezogabine as immediate release (IR) tablets three times a day (TID) as add-on therapy. Six dose strengths (25 milligrams(mg)/50 mg/100 mg/200 mg/300 mg/400 mg) were used. Doses may have been titrated no more frequently than once per week. Par. dose was adjusted as needed (e.g. based on: weight change due to increasing age and growth, efficacy or tolerability). Maximum doses allowed in the study were 900 mg per day (mg/day) (>50 kilogram (kg) weight) or 450 mg/day (30 to 50 kg weight) for par. aged <16 years old and the maximum doses allowed were 1200 mg/day (>50 kg weight) or 600 mg/day (30 to 50 kg weight) for par. aged >=16 years old.
Period: Overall Study
Arm/Group | Retigabine/Ezogabine TID
Started | 4
Completed | 0
Not Completed | 4
Not completed — Study Closed/Terminated | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Retigabine/Ezogabine TID: Par. received retigabine/ezogabine as IR tablets TID as add-on therapy. Six dose strengths (25 mg/50 mg/100 mg/200 mg/300 mg/400 mg) were used. Doses may have been titrated no more frequently than once per week. Par. dose was adjusted as needed (e.g. based on: weight change due to increasing age and growth, efficacy or tolerability). Maximum doses allowed in the study were 900 mg/day (>50 kilogram (kg) weight) or 450 mg/day (30 to 50 kg weight) for par. aged <16 years old and the maximum doses allowed were 1200 mg/day (>50 kg weight) or 600 mg/day (30 to 50 kg weight) for par. aged >=16 years old.
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.3 (1.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  White/Caucasian/European Heritage | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Par.) With Any Adverse Event (AE) or Serious Adverse Event (SAE) During the Treatment Period
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of the study medication, whether or not considered related to the study medication. A SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability or incapacity, or is a congenital anomaly or birth defect. Medical or scientific judgment was exercised in deciding whether reporting was appropriate in other situations. Please refer to the AE/SAE module for a list of non-serious AEs and SAE.
Time Frame: From the start of study medication until the end of Follow-Up (up to 178 days)
Population: All Subjects Population: all participants who enrolled in the study.
Measure: Number; unit: Participants
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 4
Participants
  Any AE | 4
  Any SAE | 0

2. Primary Outcome: Number of Participants With AEs Leading to Withdrawal
Description: as for outcome 1
Time Frame: From the start of study medication until the end of the Follow-Up Visit (up to 178 days)
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 4
Participants | 0

3. Primary Outcome: Number of Participants With Vital Signs Outside the Pre-determined Clinically Important Findings or Outside the Normal Ranges at Any Time During the Study
Description: Vital sign assessment included systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate and body temperature measurements. SBP, DBP and heart rate were measured at the following Visits: 1, 4, 5, 6, 7, EW and the FU Visit after the participants were in the seated position for 5 minutes.
Time Frame: Eligibility Assessment (Visit 1), Visit 4, Visit 5, Visit 6, Visit 7, Early Withdrawal (EW) Visit, and Follow-Up (FU) Visit (up to 178 days)
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 4
Participants | 0

4. Primary Outcome: Change From Baseline in SBP and DBP at the Indicated Time Points
Description: Vital sign assessment included SBP and DBP measurements. SBP and DBP were measured at the following Visits: 1, 4, 5, 6, 7, EW, and the FU Visit after the participant was in seated position for 5 minutes. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: Baseline, Eligibility Assessment (Visit 1), Visit 4, Visit 5, Visit 6, Visit 7, Early Withdrawal (EW) Visit, and Follow-Up (FU) Visit (up to 178 days)
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

5. Primary Outcome: Change From Baseline in Heart Rate at the Indicated Time Points
Description: Vital sign assessment included heart rate measured at the following Visits: 1, 4, 5, 6, 7, EW, and the FU Visit after the participant was in seated position for 5 minutes. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: as for outcome 4
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

6. Primary Outcome: Change From Baseline in Body Temperature at the Indicated Time Points
Description: Vital sign assessment included body temperature measurements at the following Visits: 1, 4, 5, 6, 7, EW, and the FU Visit. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: as for outcome 4
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

7. Primary Outcome: Change From Baseline in Body Height at Indicated Time Points
Description: Body height was measured without shoes and wearing light clothing at the following Visits: 1, 4, 5, 6, 7, EW and the FU Visit. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: as for outcome 4
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

8. Primary Outcome: Change From Baseline in Body Weight at the Indicated Time Points
Description: Body weight was measured without shoes and wearing light clothing at the following Visits: 1, 4, 5, 6, 7, EW and FU Visit. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: as for outcome 4
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

9. Primary Outcome: Change From Baseline in Body Mass Index (BMI) at the Indicated Time Points
Description: BMI is calculated as weight in kilograms (kg) divided by the square of their height in metres (m^2). BMI was measured at the following Visits: 1, 4, 5, 6, 7, EW and FU Visit. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: as for outcome 4
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

10. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) at the Indicated Time Points
Description: The 12-lead ECG was recorded in a supine position at the Eligibility Assessment Visitand the EW Visit after having kept a participant at rest in this position for 10 minutes. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: Baseline, Eligibility Assessment (Visit 1), EW Visit (up to 178 days)
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

11. Primary Outcome: Number of Participants With Abnormal Clinically Significant ECG Findings Based on Investigator Judgment at Anytime During the Study
Description: The 12-lead ECG was recorded in a supine position at the Eligibility Assessment Visit andthe EW Visit after having kept a participant at rest in this position for 10 minutes. Abnormal findings were analyzed as clinically significant (CS) and not clinically significant (NCS). The study investigator judged the ECG abnormailities as CS or NCS.
Time Frame: Eligibility Assessment and EW Visit
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 4
Participants | 0

12. Primary Outcome: Change From Baseline in ALT, ALP, AST, CK, and LDH Measurements at the Indicated Time Points
Description: Clinical laboratory assessments included hematology, chemistry and urinalysis parameters. Alanine amino transferase (ALT), alkaline phosphotase (ALP), aspartate amino transferase (AST), creatine kinase (CK), and lactate dehydrogenase (LDH) parameters were measured at Visits 1, 4, 5, 6, 7, EW and the FU Visit. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: as for outcome 4
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

13. Primary Outcome: Change From Baseline in Albumin, Total Protein, Hemoglobin, and Mean Corpuscle Hemoglobin Measurements at the Indicated Time Points
Description: Clinical laboratory assessments included hematology, chemistry and urinalysis parameters. Albumin, total protein, hemoglobin, and mean corpuscle hemoglobin concentration parameters were measured at Visits 1, 4, 5, 6, 7, EW and the FU Visit. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: as for outcome 4
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

14. Primary Outcome: Change From Baseline in the BUN/Creatinine and the Urine Albumin/Creatinine Ratios at the Indicated Time Points
Description: Clinical laboratory assessments included hematology, chemistry and urinalysis parameters. Blood Urea Nitrogen (BUN)/Creatinine and Urine Albumin/Creatinine were measured at Visits 1, 4, 5, 6, 7, EW and the FU Visit. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: as for outcome 4
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

15. Primary Outcome: Change From Baseline in Calcium, Carbon Dioxide Content/Bicarbonate, Chloride, Cholesterol, Glucose, Magnesium, Inorganic Phosphorus, Potassium, Sodium, and Urea/BUN Measurements at the Indicated Time Points
Description: Clinical laboratory assessments included hematology, chemistry and urinalysis parameters. Calcium, carbon dioxide content/bicarbonate, chloride, cholesterol, glucose, magnesium, inorganic phosphorus, potassium, sodium, and urea/BUN parameters were measured at Visits 1, 4, 5, 6, 7, EW and the FU Visit. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: as for outcome 4
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

16. Primary Outcome: Change From Baseline in Creatinine, Direct Bilirubin, Indirect Bilirubin, Total Bilirubin, Uric Acid, and Urine Creatinine Concentration Measurements at the Indicated Time Points
Description: Clinical laboratory assessments included hematology, chemistry and urinalysis parameters. Creatinine, direct bilirubin, indirect bilirubin, total bilirubin, uric acid, and urine creatinine concentration parameters were measured at Visits 1, 4, 5, 6, 7, EW and the FU Visit. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: as for outcome 4
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

17. Primary Outcome: Change From Baseline in Thyroid Stimulating Hormone (TSH) and Urine Albumin Measurements at the Indicated Time Points
Description: Clinical laboratory assessments included measurements of endocrine and urinalysis parameters. TSH and urine albumin parameters were measured at Visits 1, 4, 5, 6, 7, EW and the FU Visit. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: as for outcome 4
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

18. Primary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Platelet Count, Segmented Neutrophils, Total Neutrophils, and White Blood Cell Count Measurements at the Indicated Time Points
Description: Clinical laboratory assessments included hematology, chemistry and urinalysis parameters. Basophils, eosinophils, lymphocytes, monocytes, platelet count, segmented neutrophils, total neutrophils (Total absolute neutrophil count- total ANC), and white blood cell count parameters were measured at Visits 1, 4, 5, 6, 7, EW and the FU Visit. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: as for outcome 4
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

19. Primary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Platelet Count, Segmented Neutrophils, Total Neutrophils, and Red Cell Distribution Width (RDW) Percentages at the Indicated Time Points
Description: Clinical laboratory assessments included hematology, chemistry and urinalysis parameters. Basophils, eosinophils, lymphocytes, monocytes, segmented neutrophils, total neutrophils and red cell distribution width (RDW) parameters were measured at Visits 1, 4, 5, 6, 7, EW and the FU Visit. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: as for outcome 4
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

20. Primary Outcome: Change From Baseline in the Hematocrit Measurements at the Indicated Time Points
Description: Clinical laboratory assessments included hematology, chemistry and urinalysis parameters. Hematocrit was measured at Visits 1, 4, 5, 6, 7, EW and the FU Visit. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: as for outcome 4
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

21. Primary Outcome: Change From Baseline in the Mean Corpuscle Volume and Mean Platelet Volume Measurements at the Indicated Time Points
Description: Clinical laboratory assessments included hematology, chemistry and urinalysis parameters. Mean corpuscle volume and mean platelet colume parameters were measured at Visits 1, 4, 5, 6, 7, EW and the FU Visit. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: as for outcome 4
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

22. Primary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin at the Indicated Time Points
Description: Clinical laboratory assessments included hematology, chemistry and urinalysis parameters. Mean corpuscle hemoglobin was measured at Visits 1, 4, 5, 6, 7, EW and the FU Visit. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: as for outcome 4
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

23. Primary Outcome: Change From Baseline in the Red Blood Cell Count Measurements at the Indicated Time Points
Description: Clinical laboratory assessments included hematology, chemistry and urinalysis parameters. The red blood cell count was measured at Visits 1, 4, 5, 6, 7, EW and the FU Visit. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: as for outcome 4
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

24. Primary Outcome: Number of Partcipants With Hematology, Chemistry and Urinalysis Parameters Outside the Normal Ranges and Pre-determined Clinically Important Ranges
Description: Clinical laboratory assessment included hematology, chemistry and urinalysis parameters. Clinical laboratory parameters were measured at Visit 1, 4, 5, 6, 7, EW and FU Visit. Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: as for outcome 3
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

25. Primary Outcome: Changes From Baseline in Bladder Volume as Assessed by the Post Void Residual (PVR) Ultrasound at the Indicated Time Points
Description: The PVR urine test measured the amount of urine left in the bladder after urination. The PVR bladder ultrasound was performed by an urologist, a qualified technician or by an appropriately trained qualified study nurse at Visits 1, 6, and the EW Visit. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose values. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: Baseline, Eligibility Assessment (Visit 1), Visit 6, EW Visit
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

26. Primary Outcome: Changes From Baseline in Cognition as Measured by the Leiter-R at the Indicated Time Points
Description: he Leiter International Performance Scale or simply Leiter is an intelligence test for children and adolescents, with norms ranging from 2 to 20 years. For all ages, it yields an intelligence quotient (IQ) and a measure of logical ability. It is comprised of ten subtests, seven of which were relevant to the 12-18 years age group. The administration time was approximately 40 minutes. During the study, only the parent/caregiver completed this questionnaire while the participants were within the age range (i.e. <20 years). Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). The parent study did not measure baseline cognition, behavior, and learning so changes from baseline were not available for participants in this study.
Time Frame: Baseline, Eligibility Assessment (Visit 1) up to 178 days
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

27. Primary Outcome: Changes From Baseline in Behaviour as Measured by the Child Behavior Checklist (CBCL) at the Indicated Time Points
Description: The CBCL is a widely used parent report questionnaire identifying behavioural and emotional problems in children. The checklist is comprised of a number of statements about the child's behavior, e.g. acts too young for his/her age. Responses were recorded on a likert scale: 0 = not true, 1 = somewhat or sometimes true, 2 = very true or often true. The preschool checklist contained 100 questions and the school-age checklist contained 120 questions. During the study, only the parent/caregiver completed this questionnaire while the participants were within the age range (i.e. <18 years). Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). The parent study did not measure baseline cognition, behavior, and learning so changes from baseline were not available for participants in this study.
Time Frame: Baseline, Eligibility Assessment (Visit 1) up to 178 days
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

28. Primary Outcome: Changes From Baseline in Learning as Measured by the Wide Range Assessment of Memory and Learning , 2nd Edition (WRAML2) at the Indicated Time Points
Description: The WRAML2 is a standardized test that measures an individual's memory functioning. It evaluates both visual and verbal, immediate and delayed memory ability along with the acquisition of new learning. The WRAML2 core battery is composed of two verbal, two visual, and two attention concentration subtests, yielding a verbal memory index, a visual memory index and an attention-concentration index. Together, these tests yield the general memory index. The administration time is approximately 40 minutes. During the study, this test was administered if the participant was within the age range (i.e. >9 years). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). The parent study did not measure Baseline cognition, behavior, and learning so changes from Baseline were not available for participants in this study.
Time Frame: Baseline, Eligibility Assessment (Visit 1) up to 178 days
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

29. Primary Outcome: Number of Participants With Sexual Maturation Based on the Tanner Stage I to Stage V of Puberty in Participants <=18 Years Old Throughout the Study
Description: The number of participants who advanced a stage between the eligibility visit and the EW Visit was recorded. Tanner stage I is defined as no pubic hair at all (prepubertal Dominic state); stage II is defined as a small amount of long, downy hair with slight pigmentation at the base of the penis and scrotum (males) or on the labia majora (females); stage III is defined as when the hair becomes more coarse and curly, and begins to extend laterally; stage IV is defined as adult-like hair quality, extending across pubis but sparing medial thighs; and stage V is defined as when the: hair extends to medial surface of the thighs. The investigator assessed the participant's sexual development in participants <18 years old based on the Tanner Stages of Puberty.
Time Frame: Eligibility Assessment (Visit 1) and EW Visit
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 4
Participants
  Stage I to Stage II | 0
  Stage II to Stage III | 0
  Stage III to Stage IV | 0
  Stage IV to Stage V | 2
  Stage V | 2

30. Primary Outcome: Number of Days of Exposure to Retigabine/Ezogabine TID by Individual Participant
Description: Total number of days each participant was exposed to Retigabine/Ezogabine are recorded here.
Time Frame: Treatment Phase plus Taper Phase (up to 97 days)
Population: All Subjects Population
Measure: Number; unit: Days
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 4
Days
  Participant 1 | 133
  Participant 2 | 213
  Participant 3 | 196
  Participant 4 | 166

31. Secondary Outcome: Percent Change From Baseline in the Seizure Frequency at the Indicated Time Points
Description: The percentage reduction from Baseline in the seizure frequency was summarized using descriptive statistics. The frequencies and percentages were computed for a reduction in seizure frequency of >50% as well as for a 100% reduction (seizure-free). Increases of >50% in seizure frequency was also summarized. The percentage of seizure-free days wasere also analyzed. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: Basline, Eligibility Assessment (Visit 1) up to 178 days
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

32. Secondary Outcome: Number of Participants Who Were Responders During the Treatment Period
Description: A ''responder'' is defined as >50% reduction from Baseline in the seizure frequency. Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: Eligibility Assessment (Visit 1) up to 178 days
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

33. Secondary Outcome: Clinical Global Impression- Improvement (CGI-I) Assessment at the Indicated Time Points
Description: The Clinical Global Impression (CGI) scale provided an overall clinician-determined summary measure. It had 2 components: the CGI-Severity of Illness (CGI-S) scale and the CGI- Improvement (CGI-I) scale which rated the change from Baseline. The CGI-I scale scores range from 0 to 7 and are interpreted as 0=not assessed, 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: Baseline, Eligibility Assessment (Visit 1) up to 178 days
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

34. Secondary Outcome: Clinical Global Impression-Severity of Illness (CGI-S) Assessment at the Indicated Time Points
Description: The Clinical Global Impression (CGI) scale provided an overall clinician-determined summary measure. It had 2 components: the CGI-Severity of Illness (CGI-S) scale and the CGI-Improvement (CGI-I) scale which rated the change from Baseline. The CGI-S was a 7-point scale that required the investigator to rate the severity of the participant's epilepsy relative to the investigator's past experience with other participants with the same diagnosis. The CGI-S scale scores range from 0 to 7 and are interpreted as 0=not assessed, 1=normal, 2=borderline, 3=mild, 4=moderate, 5=marked, 6=severe, 7=extremely severe. Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: Baseline, Eligibility Assessment (Visit 1) up to 178 days
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

35. Secondary Outcome: Change From Baseline in Child Health Status as Measured by the Child Health Questionnaire (CHQ) in Participants <18 Years Old at the Indicated Time Points
Description: The CHQ comprises scales specifically developed for children and adolescents aged five years and older. The CHQ assesses a child's physical, emotional, and social well-being from the perspective of a parent or guardian. The questionnaire was completed by a parent/caregiver and administration time was approximately 30 minutes. The parent/caregiver completed this questionnaire while the participant was within the age range (i.e. <18 years). Baseline was the first pre-Retigabine assessment conducted in the parent study GSK113284 (NCT014945840). Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: Baseline, Eligibilty Assessment (Visit 1), EW Visit and FU Visit (up to 178 days)
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

36. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC) Following Oral Administration of Retigabine/Ezogabine at the Indicated Time Points
Description: AUC is defined as the area under the plasma drug concentration-time curve, reflects the actual body exposure to drug after administration of a dose of the drug and is expressed in milligram*hour per Liter (mg*h/L). Blood samples for population PK analysis of retigabine/ezogabine were taken at clinic visits where routine clinical laboratory samples were also taken. Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled.
Time Frame: Eligibility Assessment (Visit 1) up to 178 days
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

37. Secondary Outcome: Apparent Clearance (CL/F) Following Oral Administration of Retigabine/Ezogabine at Indicated Time Points
Description: Blood samples for population pharmacokinetic analysis of retigabine/ezogabine were taken at clinic visits where routine clinical laboratory samples were also taken. CL/F, where CL is the calculated as dose/AUC and F is the oral bioavailability of the drug. Because the study was terminated prematurely and the sample size is small, summary statistics were not compiled
Time Frame: Eligbility Assessment (Visit 1), up to 178 days
Population: All Subjects Population
Arm/Group | Retigabine/Ezogabine TID
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Non-serious adverse event (AE) and serious adverse events (SAE) were collected from the start of study treatment until the Follow-Up contact (Up to 178 days)
Description: SAEs and non-serious AEs are reported for members of the Safety Population, comprised of participants who took at least one dose of investigational product after being enrolled into the study.
Groups:
- Retigabine/Ezogabine TID: Par. received retigabine/ezogabine as IR tablets TID as add-on therapy. Six dose strengths (25 mg/50 mg/100 mg/200 mg/300 mg/400 mg) were used. Doses may have been titrated no more frequently than once per week. Par. dose was adjusted as needed (e.g. based on: weight change due to increasing age and growth, efficacy or tolerability) over the course of this long-term open-label extension study. Physicians used their clinical judgment in making dose adjustments. Maximum doses allowed in the study were 900 mg/day (>50 kilogram (kg) weight) or 450 mg/day (30 to 50 kg weight) for par. aged <16 years old and the maximum doses allowed were 1200 mg/day (>50 kg weight) or 600 mg/day (30 to 50 kg weight) for par. aged >=16 years old.
Arm/Group | Retigabine/Ezogabine TID
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Retigabine/Ezogabine TID (N=4)
Vomiting (Gastrointestinal disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Migraine (Nervous system disorders) | 1
Viral infection (Infections and infestations) | 1
Pyrexia (General disorders) | 1
Headache (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
This study was terminated early and only 4 of the planned 500 participants were enrolled. Due to the early study termination and small sample size, many planned analyses were not completed therefore lmiited results data were available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.